CLINICAL TRIAL: NCT02483377
Title: Breast Cancer Patient Navigation and Tailored Treatment Planning: A Process Evaluation Study for LAC+USC Patient Navigation, Treatment Planning, and Ongoing Support for Latina Women
Brief Title: Patient Navigation and Tailored Treatment Planning in Latina Patients With Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1B-14-7; NCI-2015-00351 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-14-7 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Breast Carcinoma
Keywords: Sign or Symptom
MeSH Terms: conditions — Breast Neoplasms; Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (treatment summaries and plan report): Patients receive treatment summaries and plan report that captures patient data through the use of an "intake checklist" completed during the initial consultation with the breast oncology team and used to guide referrals to existing services and programmed with generic information related to disease and treatment management plan. Additional elements, such as psycho-social services, exercise, and/or nutrition, identified by the patient self-report, will be incorporated. Patients also complete 3 questionnaires at each clinic visit.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This research trial studies how well patient navigation and tailored treatment planning work in Latina patients with breast cancer. Patient navigation and tailored treatment planning may provide extra support by guiding patients through the healthcare system, remove barriers to care and provide ease of access to essential resources, encourage patient participation in their care, provide in-language summaries and plans for follow-up care, improve patient access to needed supportive care services and may improve general healthcare experience in Latina patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Successful navigation of patients being screened or treated for breast cancer through the continuum of their care (from visit to visit; from surgical care to radiologic care to oncologic care; from oncologic care to supportive care; etc).

II. Supply individualized in-language treatment summaries and follow-up care plans to enrolled patients.

III. Supply tailored in-language survivorship plan summaries to enrolled patients.

OUTLINE:

Patients receive treatment summaries and plan report that captures patient data through the use of an "intake checklist" completed during the initial consultation with the breast oncology team and used to guide referrals to existing services and programmed with generic information related to disease and treatment management plan. Additional elements, such as psycho-social services, exercise, and/or nutrition, identified by the patient self-report, will be incorporated. Patients also complete 3 questionnaires at each clinic visit.

After completion of study, patients are followed up at 6 months or 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving ongoing care at LAC+USC
* Self-identified as Latina (or Hispanic)
* Known or suspected breast cancer
* Being seen in a breast cancer high risk, screening or prevention program or clinic or in one of the breast cancer clinics (surgical or medical oncology)

Exclusion Criteria:

* Inability to sign informed consent or complete questionnaires and forms
* Self-identified as non-Latina (or non-Hispanic)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Self-identified Latina (or Hispanic) who is receiving ongoing care at LAC+USC Medical Center will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Number of missed appointments from the time of initial diagnosis to the completion of primary treatment (chemotherapy, surgery and radiation as applicable) as measured by CCCQ | Up to 12 months
  Questionnaire scores will be expressed as median values with 95% confidence intervals.
Number of patients enrolled on clinical trials (interventional and non-interventional) | Up to 12 months
  Number of patients enrolled on clinical trials (interventional and non-interventional) will be quantified and compared to historical controls.
Number of special referrals made | Up to 12 months
  Number of special referrals made (eg. social worker, genetic counseling, fertility) through the navigation system will quantified and compared to historical controls.
Overall experience with breast cancer (broadly) and at LAC+USC as measured by experience-based questionnaire | Up to 12 months
Usefulness, accessibility, and quality of the patient navigation model as measured by Continuity/Coordination of Care Questionnaire (CCCQ) | Up to 12 months
  Means and standard deviations will be summarized per outcome measures at 3, 6, and 12 months after baseline, and 95% confidence intervals for the difference in means will be calculated for each assessment time for total scores and subscale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Macdonald, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States